CLINICAL TRIAL: NCT07351058
Title: A Phase III, Randomized, Double-Blind, Placebo-Controlled, Parallel Group Study to Evaluate the Efficacy and Safety of Once-Weekly RO7795068 Administered to Participants With Obesity or Overweight and Type 2 Diabetes
Brief Title: A Clinical Study to Evaluate the Effects of RO7795068 in Participants With Obesity or Overweight and Type 2 Diabetes
Acronym: Enith2
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: WC45726; 2025-523106-32-00 (EU CTIS Number)
Record Dates: First submitted 2026-01-16; First posted 2026-01-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Obesity or Overweight; Type 2 Diabetes Mellitus
MeSH Terms: conditions — Obesity; Overweight; Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Arm 1: Placebo (Placebo Comparator)
  Interventions: Combination Product: Placebo
- Arm 2: RO7795068 Dosing Regimen 1 (Experimental)
  Interventions: Combination Product: RO7795068
- Arm 3: RO7795068 Dosing Regimen 2 (Experimental)
  Interventions: Combination Product: RO7795068
- Arm 4: RO7795068 Dosing Regimen 3 (Experimental)
  Interventions: Combination Product: RO7795068

INTERVENTIONS:
Combination Product: Placebo — Placebo will be volume-matched and administered once weekly using an integrated drug-device combination product.
  Arms: Arm 1: Placebo
Combination Product: RO7795068 — RO7795068 will be administered once weekly at the randomized dosing regimen using an integrated drug-device combination product.
  Other Names: CT-388; RG6640
  Arms: Arm 2: RO7795068 Dosing Regimen 1; Arm 3: RO7795068 Dosing Regimen 2; Arm 4: RO7795068 Dosing Regimen 3

SUMMARY:
The purpose of this study is to assess the efficacy and safety of RO7795068, a dual glucagon-like peptide-1 (GLP-1)/glucose-dependent insulinotropic polypeptide (GIP) receptor agonist (RA), at multiple doses compared with placebo for weight management in participants with obesity or overweight and Type 2 diabetes mellitus (T2DM).

ELIGIBILITY:
Inclusion Criteria:

* Ability and willingness to self-administer the study drug (or receive an injection from a trained individual if visually impaired or with physical limitations)
* Diagnosis of type 2 diabetes mellitus (T2DM) according to WHO classification or other locally applicable standards with HbA1c ≥6.5% to ≤10% determined by laboratory test at screening, and on stable oral therapy for at least 3 months prior to screening (if applicable). T2DM may be treated with diet/exercise alone or any oral anti-hyperglycemic medication (as per local labeling) EXCEPT dipeptidyl peptidase 4 (DPP-4) inhibitors or GLP-1 RA-based therapy.
* Body mass index (BMI) ≥27.0 kg/m^2
* History of ≥1 self-reported unsuccessful diet/exercise effort to lose body weight

Exclusion Criteria:

* History of type 1 diabetes mellitus (T1DM) or any lifetime history of ketoacidosis or history of hyperosmolar state/coma within 12 months prior to screening
* Have had 1 or more episodes of severe hypoglycemia and/or has hypoglycemia unawareness within the 6 months prior to screening
* At least 2 confirmed fasting blood glucose values >270 mg/dL (15.0 mmol/L) (on 2 non-consecutive days) during screening
* Self-reported change in body weight >5 kg within 3 months prior to screening
* Obesity induced by other endocrinologic disorders (e.g., Cushing's syndrome) or diagnosed monogenetic or syndromic forms of obesity (e.g., melanocortin 4 receptor deficiency or Prader-Willi syndrome)
* Prior or planned surgical treatment for obesity. Liposuction or abdominoplasty if performed more than 1 year prior to screening is allowed.
* Known clinically significant gastric emptying abnormality (e.g., severe gastroparesis or gastric outlet obstruction)
* Poorly controlled hypertension at screening
* Have any of the following cardiovascular conditions within 3 months prior to screening: Acute myocardial infarction; Cerebrovascular accident (stroke)/transient ischemic attack; Unstable angina; Hospitalization due to congestive heart failure
* Treatment with any approved or investigational GLP-1-RA-based therapy (e.g., GLP-1 receptor mono agonist, GLP-1/GIP receptor dual agonist, GLP-1/GIP/Gluc receptor triple agonist) within 6 months prior to randomization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1600 (Estimated)
Dates: Start 2026-02-27 (Estimated); Primary Completion 2028-08-07 (Estimated); Study Completion 2028-08-07 (Estimated)

PRIMARY OUTCOMES:
Percent (%) Change from Baseline in Body Weight at Week 72 | Baseline through Week 72

SECONDARY OUTCOMES:
Percentage of Participants Achieving ≥5% Body Weight Loss from Baseline at Week 72 | Baseline and Week 72
Percentage of Participants Achieving ≥10% Body Weight Loss from Baseline at Week 72 | Baseline and Week 72
Percentage of Participants Achieving ≥15% Body Weight Loss from Baseline at Week 72 | Baseline and Week 72
Change from Baseline in Body Weight (kg) at Week 72 | Baseline through Week 72
Change from Baseline in Hemoglobin A1c (HbA1c) at Week 72 | Baseline through Week 72
Percentage of Participants Achieving HbA1c of ≤6.5% at Week 72 | Week 72
Percentage of Participants Achieving HbA1c of <7% at Week 72 | Week 72
Change from Baseline in Waist Circumference (cm) at Week 72 | Baseline through Week 72
Change from Baseline in Fasting Glucose at Week 72 | Baseline through Week 72
Change from Baseline in Fasting Insulin at Week 72 | Baseline through Week 72
Change from Baseline in Low-Density Lipoprotein (LDL) Cholesterol at Week 72 | Baseline through Week 72
Change from Baseline in High-Density Lipoprotein (HDL) Cholesterol at Week 72 | Baseline through Week 72
Change from Baseline in Triglyceride at Week 72 | Baseline through Week 72
Change from Baseline in Systolic Blood Pressure at Week 72 | Baseline through Week 72
Change from Baseline in the Physical Functioning Domain Score of the Short Form (36) Health Survey Version 2 (SF-36v2) Acute Form at Week 72 | Baseline through Week 72
Change from Baseline in Physical Functioning Composite Score of the Impact of Weight on Quality of Life-Lite Clinical Trials Version (IWQoL-Lite-CT) Questionnaire at Week 72 | Baseline through Week 72
Change from Baseline in Waist-to-Hip Ratio at Week 72 | Baseline through Week 72
Change from Baseline in Waist-to-Height Ratio at Week 72 | Baseline through Week 72
Change from Baseline in Subscale Scores of the Control of Eating Questionnaire (CoEQ) at Week 72 | Baseline through Week 72
Change from Baseline in Symptoms and Impact of Urinary Incontinence as Assessed by the International Consultation on Incontinence Questionnaire-Urinary Incontinence Short Form (ICIQ-UI SF) at Week 72 | Baseline through Week 72
Percentage of Participants Experiencing No Change, Improvement, or Worsening on the Patient Global Impression of Change (PGI-C) Urinary Incontinence Questionnaire at Week 72 | Baseline and Week 72
Percentage of Participants Experiencing No Change, Improvement, or Worsening on the Patient Global Impression of Severity (PGI-S) Urinary Incontinence Questionnaire at Week 72 | Baseline and Week 72
Percentage of Participants Experiencing No Change, Improvement, or Worsening on the PGI-C Physical Functioning Questionnaire at Week 72 | Baseline and Week 72
Percentage of Participants Experiencing No Change, Improvement, or Worsening on the PGI-S Physical Functioning Questionnaire at Week 72 | Baseline and Week 72
Change from Baseline in Health-Related Quality of Life (HRQoL) as Assessed by the SF-36v2 Acute Form Domain Scores and Component Summary Scores at Week 72 | Baseline through Week 72
Change from Baseline in HRQoL as Assessed by the IWQoL-Lite-CT Domain Scores and Total Score at Week 72 | Baseline through Week 72
Change from Baseline in Non-HDL Cholesterol at Week 72 | Baseline through Week 72
Change from Baseline in VLDL Cholesterol at Week 72 | Baseline through Week 72
Change from Baseline in Total Cholesterol at Week 72 | Baseline through Week 72
Change from Baseline in Free Fatty Acids at Week 72 | Baseline through Week 72
Change from Baseline in Diastolic Blood Pressure at Week 72 | Baseline through Week 72
Change from Baseline in High-Sensitivity C-reactive Protein (hsCRP) at Week 72 | Baseline through Week 72
Change from Baseline in Urinary Albumin/Creatinine Ratio at Week 72 | Baseline through Week 72
Change from Baseline in Body Mass Index (BMI) at Week 72 | Baseline through Week 72
Percent (%) Change from Baseline in Body Weight by Obesity Class at Week 72 | Baseline through Week 72
Time to Achieve ≥5%, ≥10%, or ≥15% Body Weight Loss from Baseline Through Week 72 | From Baseline through Week 72
Percentage of Participants Achieving HbA1c of <5.7% at Week 72 | Week 72
Incidence and Severity of Adverse Events, with Severity Determined According to Mild/Moderate/Severe Criteria | Baseline through Week 72
Change from Baseline in the Columbia-Suicide Severity Rating Scale (C-SSRS) Score Through Week 72 | Baseline through Week 72
Change from Baseline in the Patient Health Questionnaire-9 (PHQ-9) Score Through Week 72 | Baseline through Week 72

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche

IPD SHARING:
Plan to Share IPD: Yes
For eligible studies, qualified researchers may request access to individual patient level clinical data. See Roche's commitment to transparency of clinical study information here: https://go.roche.com/data_sharing